CLINICAL TRIAL: NCT07174908
Title: A Phase 3 Multicenter, Randomized, Controlled, and Open-Label Study of IN10018 in Combination With D-1553 Versus Standard Therapy for the Treatment of First Line Locally-advanced or Metastatic Non-squamous Non-small Cell Lung Cancer With KRAS G12C Mutation
Brief Title: A Phase 3 Study of IN10018 in Combination With D-1553 Versus Standard Therapy for First Line Non-squamous Non-small Cell Lung Cancer With KRAS G12C Mutation
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: InxMed (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IN10018-023
Record Dates: First submitted 2025-08-29; First posted 2025-09-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-09

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Platinum; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IN10018 plus D-1553 (Experimental): Subjects receive IN10018 100mg orally once daily (QD) and D-1553 600mg orally twice daily (BID) on Days 1-21 of each 21-day cycle, until disease progression or unacceptable toxicity.
  Interventions: Drug: IN10018 in combination with D-1553
- Tislelizumab plus Platinum and Pemetrexed (Active Comparator): Subjects receive Tislelizumab 200mg intravenously (IV) once every 3 weeks (Q3W) until disease progression, plus Carboplatin (AUC = 5 mg/mL/min, Q3W, IV) or Cisplatin (75 mg/m², Q3W, IV) for up to 4 cycles, in combination with Pemetrexed (500 mg/m², Q3W, IV) until disease progression.
  Interventions: Drug: anti-PD-1 monoclonal antibody in combination with platinum and pemetrexed

INTERVENTIONS:
Drug: IN10018 in combination with D-1553 — IN10018 100mg QD PO and D-1553 600mg BID PO, 21days per cycle
  Arms: IN10018 plus D-1553
Drug: anti-PD-1 monoclonal antibody in combination with platinum and pemetrexed — Tislelizumab 200mg Q3W IV + Carboplatin AUC 5 mg/mL/min or Cisplatin 75mg/m² Q3W IV+ Pemetrexed 500mg/m² Q3W IV
  Arms: Tislelizumab plus Platinum and Pemetrexed

SUMMARY:
This is a multicenter, randomized, open-label, phase III clinical study, to evaluate the efficacy and safety of IN10018 in combination with D-1553 as compared to anti-PD-1 monoclonal antibody (mAb) in combination with platinum and pemetrexed as the first-line treatment for the locally advanced or metastatic KRASG12C mutation-positive non-squamous non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
Preclinical studies indicate that IN10018 synergizes with D-1553 to enhance antitumor activity and delay resistance through multiple mechanisms, including suppression of FAK-YAP signaling pathway activation, reduction of tumor stromal fibrosis, and induction of immunogenic cell death (ICD). IN10018-602/D1553-106 is an ongoing Phase Ib/II clinical study evaluating the synergistic antitumor activity and safety of IN10018 combined with D-1553 in patients with KRAS G12C-mutant solid tumors. Preliminary results have demonstrated notable antitumor activity and a favorable safety and tolerability profile in patients with advanced KRAS G12C-mutant NSCLC and metastatic colorectal cancer. Based on the available clinical data, the sponsor plans to initiate a Phase III study in previously untreated patients with advanced KRAS G12C-mutant NSCLC to further evaluate the efficacy and safety of IN10018 in combination with D-1553 compared with first-line standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide informed consent and comply with study requirements
* Has histologically confirmed locally advanced (Stage IIIB/C) or metastatic (Stage IV) non-squamous NSCLC
* Aged 18-80 years at the time of consent
* Has KRAS G12C mutation confirmed by central laboratory
* Has not received prior systemic therapy for advanced or metastatic NSCLC
* Has at least one measurable lesion per RECIST v1.1
* ECOG performance status of 0-1
* Has adequate organ function
* Life expectancy ≥3 months in the opinion of the Investigator
* Male and female subjects of reproductive potential must agree to use effective contraception during and for 6 months after treatment

Exclusion Criteria:

* Has other histological subtypes of NSCLC (e.g., small cell or neuroendocrine)
* Has active or untreated CNS metastases or carcinomatous meningitis
* Prior treatment with KRAS G12C inhibitors, FAK inhibitors, or immune checkpoint inhibitors
* Has another known driver mutation with approved targeted therapy (e.g., EGFR, ALK, ROS1)
* Has uncontrolled cardiovascular disease, active severe infection, interstitial lung disease, or autoimmune disease requiring systemic therapy
* Has history of another malignancy within 5 years, except those curatively treated and considered low risk (e.g., basal cell carcinoma, cervical carcinoma in situ)
* Has gastrointestinal conditions that may interfere with absorption of oral drugs (if applicable)
* Has known active hepatitis B, hepatitis C, or HIV infection
* Has received a live vaccine within 30 days before first dose of study drug
* Pregnant or breastfeeding women
* Has psychiatric or substance abuse disorders that would interfere with study compliance
* Is participating in another interventional clinical study
* Any condition that, in the opinion of the Investigator, would interfere with participation or study results

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | up to 36 months
  Defined as time from randomization until disease progression or death from any cause, whichever occurs first assessed per RECIST v1.1 by blinded independent central review (BICR).

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | up to 36 months
  Defined as complete response (PR) + partial response (PR) assessed per RECIST v1.1 by BICR
Overall Survival (OS) | up to 60 months
  Defined as time from randomization to death by any cause
Disease Control Rate (DCR) | Up to 36 months
  Defined as ORR + stable disease (SD) assessed per RECIST v1.1 by BICR
Duration of Response (DoR) | up to 36 months
  Defined as time from first evidence of PR or CR to disease progression or death due to any cause, whichever occurs first. assessed per RECIST v1.1 by BICR
PFS | up to 36 months
  Defined as time from randomization until disease progression or death from any cause, whichever occurs first assessed per RECIST v1.1 by investigator assessment.
ORR | up to 36 months
  defined as CR+PR assessed per RECIST v1.1 by investigators
DCR | up to 36 months
  Defined as ORR + stable disease (SD) assessed per RECIST v1.1 by investigators
DOR | Up to 36 months
  Defined as time from first evidence of PR or CR to disease progression or death due to any cause, whichever occurs first. assessed per RECIST v1.1 by investigators
Number of subjects with adverse event | up to 36 months
  The number of subjects who experienced AEs is presented

OTHER OUTCOMES:
PK: Cmax of IN10018 and D-1553 | up to 36 months
  Maximum concentration (Cmax)
PK: Cmin of IN10018 and D-1553 | up to 36 months
  Minimum concentration (Cmin)
PK: AUC of IN10018 and D-1553 | up to 36 months
  Area under the concentration-time curve (AUC)
Patient-reported outcome (PRO) questionnaire | up to 36 months
  Reports of health status directly from patients

CONTACTS AND LOCATIONS:
Overall Officials: Zhengbo Song Professor, Doctor, Principal Investigator — Zhejiang Cancer Hospital; Shun Lu Professor, Doctor, Principal Investigator — Shanghai Chest Hospital
Locations (11):
- China (11):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital Tongji Medidcal College Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - First Affiliated Hospital of Gannan Medical University, Gannan, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No